CLINICAL TRIAL: NCT04194918
Title: A Scalable E-Health Smoking Cessation Intervention for Sexual and Gender Minority Young Adults
Brief Title: Flexiquit+: Web Program to Promote Smoking Cessation in Sexual and Gender Minority Young Adult Smokers
Acronym: EQQUAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Safeway Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1004771; NCI-2019-08031 (Registry Identifier: NCI / CTRP); P30CA015704 (NIH); 10396 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (Flexiquit+, text message, handout) (Experimental): Individuals will be recruited to use the Flexiquit+ program consisting of 6 sessions, each lasting approximately 25 minutes. Participants will also receive text messages providing motivational messages and review information discussed in the program. At the end of the intervention, participants will receive an email with all of the session handouts.
  Interventions: Behavioral: Computer-Assisted Smoking Cessation Intervention; Other: Text Message; Other: Handout; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Behavioral: Computer-Assisted Smoking Cessation Intervention — Use the Flexiquit+ program
Other: Text Message — Receive text messages
  Other Names: SMS Text; SMS Text Message; Text
Other: Handout — Receive handouts via email
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial studies how well Flexiquit+ helps young adult smokers who identify as a sexual and/or gender minority to quit or cut down on smoking. Flexiquit+ is an avatar-led, web-based intervention that can help smokers quit or cut back on how much they smoke cigarettes and/or vape, reducing their chances of developing tobacco-related health conditions.

DETAILED DESCRIPTION:
OUTLINE:

Individuals will be recruited to use the Flexiquit+ program consisting of 6 sessions, each lasting approximately 25 minutes. Participants will also receive text messages providing motivational messages and review information discussed in the program. At the end of the intervention, participants will receive an email with all of the session handouts.

Participants are followed up with at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-identify as a sexual and/or gender minority (i.e., a sexual orientation other than straight and/or gender that doesn't match sex assigned at birth)
* Participants must currently reside in the United States and anticipate remaining in the United States for the duration of the study (2 months)
* Participants must self-report smoking at least 1 cigarette per day in the 30 days prior to screening
* Participants must self-report having at least weekly internet access for the next two months
* Participants must self-report being willing and able to stream video online for this study
* Participants must self-report current use of a personal email account
* Participants must self-report current use of text messaging
* Participants must self-report that they are interested in participating in the study for themselves (versus [vs] someone else)
* Participants must self-report that they are not currently taking part in any other smoking cessation treatment such as the nicotine patch, nicotine gum, Zyban, in-person counseling, telephone counseling, using a web-based or app-based cessation program
* Participants must self-report that they have not participated in one of our prior smoking cessation studies, including the user-centered research conducted in the development of Flexiquit+
* Participants must self-report that they are comfortable reading, writing, and speaking English
* Participants must self-report that they understand and agree to the conditions of compensation
* Participants must self-report that they are not currently incarcerated in a prison
* Participants must be willing to use the Flexiquit+ program, complete the study assessments, and sign an online consent form

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Treatment utilization | Enrollment up to 2 months
  Will be determined by the server-recorded number of logins and the number of sessions completed. Frequencies (for categorical variables) or means and standard deviations (for continuous variables) will be reported for treatment utilization and satisfaction. Tables with N (%) or mean (standard deviation) by treatment arm will be provided.
Treatment satisfaction: survey | Enrollment up to 2 months
  Will be determined using 12 items on the 2-month outcome survey. Frequencies (for categorical variables) or means and standard deviations (for continuous variables) will be reported for treatment utilization and satisfaction. Categorical ratings for treatment satisfaction questions will be dichotomized as "somewhat", "mostly", or "very" useful versus (vs.) lower ratings. Tables with N (%) or mean (standard deviation) by treatment arm will be provided.

SECONDARY OUTCOMES:
Smoking cessation rate | At 2 months post-enrollment
  Will be assessed using the self-reported 7-day point prevalence abstinence at 2-month follow-up survey, biochemically confirmed with saliva cotinine.
Change in motivation to quit smoking | From baseline to 2-month follow-up
  Will be assessed using the Contemplation Ladder.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT04194918/ICF_000.pdf